CLINICAL TRIAL: NCT04602299
Title: Setting the Shortest Examination Time of Gastroscopy to Improve the Detection Rate of Upper Gastrointestinal Tumors: a Multi-center, Prospective, Controlled Study
Brief Title: Setting the Shortest Examination Time of Gastroscopy to Improve the Detection Rate of Upper Gastrointestinal Tumors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Zhaoshen Li, Director of Gastroenterology, Changhai Hospital
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Screening
Other Study IDs: gastroscopy time
Record Dates: First submitted 2020-10-20; First posted 2020-10-26 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: Gastroscopy Time; Early Gastric Cancer; Detection Rate
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Set the minimum time of gastroscopy (Experimental)
  Interventions: Other: Set the minimum time of gastroscopy
- Observe the procedure time of gastroscopy (No Intervention)

INTERVENTIONS:
Other: Set the minimum time of gastroscopy — This study contains 2 stages. At the first stage, no interventions are implemented. The researchers just observe the actual procedure time of gastroscopy. At the second stage, a minimal procedure time is set based on the observational results of the first stage.
  Arms: Set the minimum time of gastroscopy

SUMMARY:
This multicenter, prospective, interventional study aims to include 2000 gastroscopic procedures and investigate the relationship between procedure time and lesion detection rate in tertiary endoscopic centers in China. At the first stage, the researchers observe the actual procedure time of gastroscopies without affecting the natural behavior of endoscopists. At the second stage, a minimal time limit will be set for each procedure based on the observational results of the first stage. The primary study outcome is focal lesion detection rate. Secondary outcomes include detection rate of early upper GI cancer, biopsy rate and adverse event rate.

DETAILED DESCRIPTION:
China is a country with a heavy burden of gastric cancer and esophageal cancer. In 2015, the incidence/mortality of gastric cancer and esophageal cancer in China were 680000/500000 and 220000/200000, respectively. Gastroscopy is the most important means to detect early cancer of gastrointestinal tract. However, due to various factors, the miss rate of clinical significant lesions by gastroscopy is innegligible. Our previous research results showed that the detection rate of early gastric cancer and early esophageal cancer in China was only about 15%. This study aims to include 2000 gastroscopic procedures and investigate the relationship between procedure time and lesion detection rate in tertiary endoscopic centers in China.

At the first stage, the researchers observe the actual procedure time of gastroscopies without affecting the natural behavior of endoscopists. Then, researchers collect the data (including focal lesion detection rate, procedure time, detection rate of early upper GI cancer, biopsy rate and adverse event rate) and analyze the minimal procedure time. At the second stage, a minimal time limit will be set for each procedure. Every stage last two months, and potential correlations between lesion detection rate and procedure time will be investigated through subsequent statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* No history of benign and malignant tumors (including carcinoma and adenoma) of upper GI (including esophagus, stomach and duodenum)
* undergo gastroscopy with intravenous anesthesia (or conscious sedation)

Exclusion Criteria:

* Subjects with focal lesions detected by gastroscopy within 1 year
* Subjects that cannot stand the gastroscopy procedure or cannot cooperate with endosccopists
* Emergency endoscopy and therapeutic endoscopy
* Subjects with history of esophageal or stomach surgery or endoscopic surgery
* Pregnant
* Subjects that taking antiplatelet or anticoagulant drugs which contradicts endoscopic biopsy
* Subjects with other serious complications that affect the speed of gastroscopy
* Subjects that refuse to cooperate with data collection or sign the informed consent

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2000 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-01-15 (Actual)

PRIMARY OUTCOMES:
focal lesion detection rate | two months
  number of gastroscopy procedures that detects focal lesions divided by the number of all gastroscopy procedures

SECONDARY OUTCOMES:
detection rate of high risk lesions | two months
  number of gastroscopy procedures that detect upper GI cancers (gastric or esophageal cancer), dysplasia and intestinal metaplasia divided by the number of all gastroscopy procedures
endoscopic biopsy rate | two months
  number of gastroscopy procedures with biopsy divided by the number of all gastroscopy procedures
detection rate of neoplastic lesions | two months
  number of gastroscopy procedures that detect upper GI cancers divided by the number of all gastroscopy procedures
mean (median) examination time for normal EGDs without biopsy | two months
  mean (median) examination time for all normal EGDs without biopsy
rate of procedures reaching the minimal time | two months
  number of gastroscopy procedures that reach the minimal time divided by the number of all gastroscopy procedures

CONTACTS AND LOCATIONS:
Overall Officials: Ye Gao, Principal Investigator — Changhai Hospital
Locations (2):
- China (2):
  - Changhai Hospital, Second Military Medical University, Shanghai
  - Changhai Hospital, Shanghai

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gao Y, Cai MX, Tian B, Lin H, Jiang ZY, Yang XC, Lu L, Li L, Shi LH, Liu XY, Wang YL, Li ZS, Xin L, Wang LW. Setting 6-Minute Minimal Examination Time Improves the Detection of Focal Upper Gastrointestinal Tract Lesions During Endoscopy: A Multicenter Prospective Study. Clin Transl Gastroenterol. 2023 Aug 1;14(8):e00612. doi: 10.14309/ctg.0000000000000612. PMID 37307142